CLINICAL TRIAL: NCT05417477
Title: Evaluation of a Connected Interface (Rheumatologist, Physiotherapist, Patient) to Improve the Quality of Life and the Disability of Patients With Rheumatic Diseases
Brief Title: Evaluation of a Connected Interface to Improve the Quality of Life and the Disability of Patient With Rheumatic Diseases
Acronym: RHUMATO-APP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RECHMPL21_0412
Record Dates: First submitted 2022-05-27; First posted 2022-06-14 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatic and musculoskeletal diseases; e-health; care pathway
MeSH Terms: conditions — Arthritis, Rheumatoid; Musculoskeletal Diseases

STUDY DESIGN:
Intervention Model Description: Prospective exploratory pilot study. We plan to recruit 40 patients with Chronic Inflammatory Rheumatism (CIR) and 40 patients with Osteoarthritis (OA) by several investigating teams, for a total of 80 patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- chronic inflammatory rheumatism or osteoarthritis (Experimental): The experimental intervention consists in providing the patient with access to a specific version of the application ''MedicApp'' for the duration of the study.
  The intervention will be limited for each patient to the entry of their data on the application at regular intervals during the study.
  The interface on the rheumatologist side will contain the demographic characteristics of the patient, his history, the treatments and the pathology requiring the use of physiotherapy Then, at regular intervals, the scores of the questionnaires addressed to the patient will be available on his interface. The interface, on the physiotherapist side, will contain the summary of the patient's clinical history, his treatments and the reason for the physiotherapy sessions. Then, at regular intervals, the physiotherapist will indicate the patient's locomotor assessment, the type of intervention performed and the final summary.
  Interventions: Device: use of an e-health application

INTERVENTIONS:
Device: use of an e-health application — Use of the e-health application throughout the duration of the study combined with the usual management of the disease and 20 physiotherapy sessions.

SUMMARY:
Musculoskeletal pathologies constitute a major public health problem. Rheumatologists, whether they practice in private or hospital settings, play a major role in the management of responsible for these ailments.

Due to the increase in life expectancy, an increase in the number of consultations can be expected. It is therefore imperative that the latter be more efficient, without losing quality.

Communication between doctor and patient is bound to evolve due to the multiplicity of IT tools available and those that are emerging, which are increasingly essential, including many smartphone applications. Each targeting a specific pathology (rheumatoid arthritis, ankylosing spondylitis, osteoporosis osteoarthritis, they will allow the patient to self-assess, thus becoming an actor in his own care.

A "facilitated" exchange between caregivers and patients would be relevant and would provide added value for all. This is the reason why there is a real need for an application listing precise information on the patient, in a sufficiently succinct way to optimize their transmission to the physiotherapist.

DETAILED DESCRIPTION:
Musculoskeletal pathologies constitute a major public health problem. Rheumatologists, whether they practice in private or hospital settings, play a major role in the management of responsible for these ailments.

Due to the increase in life expectancy, an increase in the number of consultations can be expected. It is therefore imperative that the latter be more efficient, without losing quality.

Communication between doctor and patient is bound to evolve due to the multiplicity of IT tools available and those that are emerging, which are increasingly essential, including many smartphone applications. Each targeting a specific pathology (rheumatoid arthritis, ankylosing spondylitis, osteoporosis osteoarthritis, they will allow the patient to self-assess, thus becoming an actor in his own care.

A "facilitated" exchange between caregivers and patients would be relevant and would provide added value for all. This is the reason why there is a real need for an application listing precise information on the patient, in a sufficiently succinct way to optimize their transmission to the physiotherapist.

Our team has recently highlighted that monitoring rheumatoid arthritis in connected mode (smartphone + online interface for the physician + distancing interaction patient / caregiver) provided a benefit in terms of quality of life as well as on the medico-economics level compared to conventional monitoring, without affecting the control of rheumatoid arthritis activity. Telemedicine is positioned more than ever as an essential instrument for organizing the longitudinal monitoring of diseases, especially in a context of confinement, which implies limited access to physiotherapy sessions, even though these are essential for optimizing the management of many osteoarticular disorders. By promoting the use of a digital telemedicine tool in the follow-up of patients suffering from rheumatological pathologies in both private practice and hospitals, the Rhumato-App project aims to develop an ergonomic offline/online platform for patients/healthcare providers (e.g. rheumatologist, general practitioner, physiotherapist), accessible from a computer or a smartphone. This platform will improve the articulation of the patient's care pathway by feeding a secure medical file shared between caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 70 years
* Presence of a chronic inflammatory rheumatism (rheumatoid arthritis, axial and/or peripheral spondyloarthritis) or osteoarthritis disease requiring the initiation of at least 20 sessions of physical therapy
* Diagnostic confirmation left to the discretion of the investigating physician
* Accessibility of an internet network (compatible with smartphone and/or computer)
* Information and consent of the patient

Exclusion Criteria:

* Pregnant or breastfeeding women
* Patient refusing or unable to give consent: patient under guardianship or curator, mentally retarded, dementia, language barrier
* Patient not affiliated to a social security scheme
* Patient under legal protection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2023-12-22 (Estimated); Study Completion 2023-12-22 (Estimated)

PRIMARY OUTCOMES:
Change of the quality of life of patients between baseline and 6 months | between baseline and 6 months
  Evaluate the impact of the computer interface on the patient's quality of life by comparing the evolution of the global SF-12 score between baseline and 6 months (longitudinal follow-up).
  The Survey Form-12 (SF-12) is a self-reported outcome measure assessing the impact of health on an individual's everyday life.
  The SF-12 is a shortened version of SF-36.
  The SF-12 have eight domains :
  1. Limitations in physical activities because of health problems.
  2. Limitations in social activities because of physical or emotional problems
  3. Limitations in usual role activities because of physical health problems
  4. Bodily pain
  5. General mental health (psychological distress and well-being)
  6. Limitations in usual role activities because of emotional problems
  7. Vitality (energy and fatigue)
  8. General health perceptions

SECONDARY OUTCOMES:
Percentage of satisfied patients | between inclusion and 6 months
  To assess the patient's satisfaction with the use of this device at the end of the 6-month follow-up with the F-SUS (French System Usability Scale) questionnaire.
  The F-SUS (French System Usability Scale) is a 10-items, to determine the level of satisfaction of users of a service and the usability of the interactive system of the study.
  Score range from 1 to 5 with 1=totally disagree and 5=totally agree
Percentage of patients adhering to the interface | between baseline and 6 months
  Evaluate the patient's adherence to the use of a computer interface based on the weekly filling rate during the 6-month follow-up
Percentage of adherent patients whose disease activity is positively impacted | between baseline and 6 months
  Assess the association between patient adherence and change in disease activity level between baseline and 6 months
Percentage of adherent patients whose quality of life is positively impacted | between baseline and 6 months
  Evaluate the association between patient compliance and the variation in their quality of life between baseline and 6 months
Percentage of adherent patients who are satisfied with the intervention | between baseline and 6 months
  Assess the association between patient adherence and satisfaction at 6 months
Percentage of satisfied caregivers | between baseline and 6 months
  Assess the satisfaction of caregivers (physiotherapist, rheumatologist) with the use of this device at the end of the 6-month follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided